CLINICAL TRIAL: NCT04513665
Title: A Phase 2 Trial of ZW25 in HER2 Overexpressed Advanced Endometrial Cancers and Carcinosarcomas (ZW25-IST-2)
Brief Title: ZW25 in Women With Endometrial Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-162
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer; Carcinosarcoma
Keywords: Endometrial Cancer; Carcinosarcoma; ZW25; 20-162; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Endometrial Neoplasms; Carcinosarcoma

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages. Stage 1 will accrue 16 patients and if two or greater responses are seen, Stage 2 will accrue an additional 9 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Experimental): Participants will have recurrent endometrial carcinoma or carcinosarcoma with HER2 overexpression and 1-2 prior lines of chemotherapy. 16 participants will be accrued. If 2 or greater responses are seen, Stage 2 will accrue additional participants.
  Interventions: Drug: ZW25
- Stage 2 (Experimental): If 2 or greater responses are seen during Stage 1, Stage 2 will accrue an additional 9 participants. Participants will have recurrent endometrial carcinoma or carcinosarcoma with HER2 overexpression and 1-2 prior lines of chemotherapy.
  Interventions: Drug: ZW25

INTERVENTIONS:
Drug: ZW25 — ZW25 at 20mg/kg intravenously (IV) every two weeks.

SUMMARY:
This study is being done to test the drug ZW25 and look at whether this drug is effective in women with HER2-overexpressed endometrial cancer or carcinosarcoma that has been treated in the past.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled or agree to consent to the companion genomic profiling study MSKCC IRB# 12-245 Part A. Results are not required prior to initiating treatment on protocol, unless patients do not have other test results by IHC or FISH confirming HER2 overexpression.
* Patients must have recurrent or persistent HER2 overexpressing endometrial cancer or endometrial carcinosarcoma. HER2 overexpression is defined as 3+ by IHC or 2+ with gene amplification by FISH (HER2/CEP17 ratio ≥ 2) or HER2 amplified (fold change ≥ 2) on MSK IMPACT.
* Histologic documentation of diagnosis of endometrial carcinoma or carcinosarcoma is required.
* Age ≥ 18 years
* Patients must have had at least one but no more than two prior chemotherapeutic regimens for management of endometrial carcinoma (including neo-adjuvant and/or adjuvant chemotherapy). Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen. Prior hormonal therapy will not count as a prior regimen. Prior treatment with trastuzumab is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* LVEF ≥ 50% on baseline screening ECHO.
* Resolution of adverse effects of recent surgery, radiotherapy, or chemotherapy to Grade ≤ 1 prior to first study treatment (with the exception of alopecia or clinically insignificant laboratory values).
* Patients must have measurable disease. Measurable disease is defined by RECIST (version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each non-nodal lesion must be 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or 20 mm when measured by chest x-ray. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.
* No active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection).
* All patients must consent to mandatory pre-treatment and post-treatment core needle biopsies.
* Patients must have adequate hematological, liver, cardiac and kidney function within 14 days prior to first treatment:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
  2. Platelet ≥ 100 X 109/L (>100,000 per mm^3)
  3. Hemoglobin ≥ 8.0 g/dL
  4. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). (Unless Gilbert's Syndrome, for which Bilirubin ≤ 3 x institutional upper limit of normal (ULN), without concurrent clinically significant liver disease) AST (SGOT)/ALT (SGPT) ≤ 3 x institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤ 5x ULN.
  5. Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN).
* For patients of childbearing potential, agreement to use two effective forms of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study and for 12 weeks after the last ZW25 dose.
* Agree to practice total abstinence when this is in line with the preferred and usual lifestyle of the subject.

  1. A woman is considered to be of childbearing potential unless 1 of the following applies: She is considered to be permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, tubal ligation, and bilateral oophorectomy.
  2. She is postmenopausal, defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 mIU/mL or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state.
  3. Female patients of childbearing potential must have a negative serum pregnancy test result less than 3 day prior to administration of the first dose of study treatment.

Patients or their legally authorized representative (LAR) must be willing and able to sign the informed consent form, and to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Women who are pregnant or lactating or women of childbearing potential (WCBP) not protected by highly-effective contraceptive methods.
* > Grade 1 peripheral neuropathy.
* History of hemorrhagic or ischemic stroke within the prior six months.
* History of NYHA Class II-IV heart failure, no serious arrhythmia.
* History of MI or unstable angina within 6 months of study initiation.
* Patients with a lifetime cumulative dose of anthracycline >300 mg/m2 or who have received anthracycline treatment within 90 days of the expected first dose of ZW25 are not eligible for treatment.
* Prior hypersensitivity to monoclonal antibodies.
* Active hepatitis B or hepatitis C infection. Patients with previously resolved hepatitis B infection are eligible. Presence of positive test results for hepatitis B infection who have resolved the infection (defined by positive for HB surface antibody (anti-HBs) and polymerase chain reaction (PCR) assay is negative for HBV DNA are eligible. Patients positive for HCV antibody are eligible only if testing for HCV RNA is negative.
* Known HIV infection.
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease).
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment.
* Known untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control) leptomeningeal carcinomatosis.

Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria:

1. Presence of measurable disease outside the CNS
2. No radiographic evidence of worsening upon the completion of CNSdirected therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
3. No history of intracranial hemorrhage or spinal cord hemorrhage
4. No ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
5. Absence of leptomeningeal disease

   * Inability to comply with study and follow-up procedures.
   * Known allergy or hypersensitivity to the components of ZW25 formulation.
   * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
   * Active or history of inflammatory bowel disease (IBD)
   * Severe infections within 4 weeks prior to initiation of study drug treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
   * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible for the study. Patients receiving antibiotic treatment for urinary tract infection are also eligible.
   * Administration of a live attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipated need for such a vaccine during study. Patients must agree not to receive live, attenuated influenza vaccine (e.g., Flumist®) within 4 weeks prior to treatment.)
   * Participation in another clinical study with receipt of an investigational product during the last 4 weeks.
   * History of another primary malignancy except for:

a. Malignancy treated with curative intent and with no known active disease ≥ 2 years before the first dose of study drug and of low potential risk for recurrence. b. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. c. Adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ). d. Adequately treated stage 1 breast cancer.

* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) < 21 days prior to the first dose of study drug. Receipt of the last dose of hormonal therapy within < 7 days prior to the first dose of study drug.
* Any prior radiation therapy must be discontinued at least four weeks prior to registration.
* QT interval corrected for heart rate (QTc) ≥ 470 ms on screening electrocardiograms (ECG) using QTC Federica.
* History of small or large bowel obstruction within 3 months of registration, including subjects with palliative gastric drainage catheters. Subjects with palliative diverting ileostomy or colostomy are allowed if they have been symptom free for more than 3 months.
* Subjects with refractory ascites, defined as ascites needing drainage catheter or therapeutic paracentesis more often than every 4 weeks.
* Ongoing bowel perforation or presence of bowel fistula or abscess within 3 months of registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikky Makker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Lumish M, Chui MH, Zhou Q, Iasonos A, Sarasohn D, Cohen S, Friedman C, Grisham R, Konner J, Kyi C, Rubinstein M, Troso-Sandoval T, Aghajanian C, Makker V. A phase 2 trial of zanidatamab in HER2-overexpressed advanced endometrial carcinoma and carcinosarcoma (ZW25-IST-2). Gynecol Oncol. 2024 Mar;182:75-81. doi: 10.1016/j.ygyno.2023.12.028. Epub 2024 Jan 22. PMID 38262242
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants accrued to Stage 2 arm.
Period: Overall Study
Arm/Group | Stage 1 | Stage 2
Started | 16 | 0
Completed | 0 | 0
Not Completed | 16 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 14 | 0

BASELINE CHARACTERISTICS:
Population: No participants accrued to Stage 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 | Stage 2 | Total
Number analyzed (Participants) | 16 | 0 | 16
Age, Continuous [Median (Full Range); unit: years] | 71 [64 to 86] |  | 71 [64 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 |  | 16
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 16 |  | 16
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 5 |  | 5
  White | 10 |  | 10
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate/ORR of Participants
Description: ORR = Compete Response (CR) + Partial Response (PR) by RECIST v 1.1 </= 24 weeks from the start of treatment
Time Frame: </= 24 weeks from the start of treatment
Population: No participants accrued to Stage 2 arm
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 | Stage 2
Number analyzed (Participants) | 16 | 0
Participants
  Participants with ORR (CR + PR) | 1 |
  Participants without ORR (CR + PR) | 15 |

ADVERSE EVENTS:
Time Frame: 24 weeks from end of treatment, up to 48 weeks
Description: No participants accrued to Stage 2 arm
Arm/Group | Stage 1 | Stage 2
All-Cause Mortality (participants affected / at risk) | 8/16 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/0
Other Adverse Events (participants affected / at risk) | 16/16 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (N=16) | Stage 2 (N=0)
Abdominal Pain (Gastrointestinal disorders) | 2 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 (N=16) | Stage 2 (N=0)
Abdominal distension (Gastrointestinal disorders) | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | NA
Allergic reaction (Immune system disorders) | 1 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | NA
Anemia (Blood and lymphatic system disorders) | 1 | NA
Anorexia (Metabolism and nutrition disorders) | 7 | NA
Ascites (Gastrointestinal disorders) | 2 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Blurred vision (Eye disorders) | 1 | NA
Catheter related infection (Infections and infestations) | 1 | NA
Colonic obstruction (Gastrointestinal disorders) | 1 | NA
Constipation (Gastrointestinal disorders) | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Diarrhea (Gastrointestinal disorders) | 12 | NA
Dry eye (Eye disorders) | 1 | NA
Dry mouth (Gastrointestinal disorders) | 1 | NA
Dysgeusia (Nervous system disorders) | 2 | NA
Dyspepsia (Gastrointestinal disorders) | 2 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Dysuria (Renal and urinary disorders) | 1 | NA
Edema limbs (General disorders) | 1 | NA
Eyebrow hair loss (Skin and subcutaneous tissue disorders) | 1 | NA
Fall (Injury, poisoning and procedural complications) | 3 | NA
Fatigue (General disorders) | 4 | NA
Fever (General disorders) | 2 | NA
Floaters (Eye disorders) | 1 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | NA
Headache (Nervous system disorders) | 1 | NA
Hemorrhoids (Gastrointestinal disorders) | 1 | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | NA
Hypertension (Vascular disorders) | 2 | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | NA
Laryngitis (Infections and infestations) | 1 | NA
Lung infection (Infections and infestations) | 1 | NA
Lymph node pain (Blood and lymphatic system disorders) | 1 | NA
Malaise (General disorders) | 1 | NA
Mucositis oral (Gastrointestinal disorders) | 1 | NA
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Nasal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Nausea (Gastrointestinal disorders) | 4 | NA
Neck edema (General disorders) | 1 | NA
Pain (General disorders) | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | NA
Palpitations (Cardiac disorders) | 2 | NA
Papulopustular rash (Infections and infestations) | 1 | NA
Paresthesia (Nervous system disorders) | 1 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | NA
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Sinus tachycardia (Cardiac disorders) | 1 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | NA
Thromboembolic event (Vascular disorders) | 1 | NA
Thrush (Infections and infestations) | 1 | NA
Upper respiratory infection (Infections and infestations) | 1 | NA
Urinary tract infection (Infections and infestations) | 1 | NA
Urinary urgency (Renal and urinary disorders) | 1 | NA
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 3 | NA
Weight loss (Investigations) | 3 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT04513665/Prot_SAP_000.pdf